CLINICAL TRIAL: NCT00257803
Title: A Randomized Double-blind Comparison of a 5 Unit Intravenous Oxytocin Bolus Versus Placebo as a Strategy to Prevent Uterine Atony at Cesarean Section in Women Who Are at Increased Risk of Post-Partum Hemorrhage
Brief Title: Does the Rapid Intravenous Administration of Oxytocin After Delivery of the Baby Decrease the Bleeding During Cesarean Section in Women at Risk of Bleeding During Cesarean Section?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H05-70504; NHR05-0206
Record Dates: First submitted 2005-11-21; First posted 2005-11-23 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-02

CONDITIONS: Postpartum Hemorrhage
Keywords: Oxytocin, bolus, postpartum hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): In the other group, the women will receive a small injection of oxytocin directly into the vein via their intravenous (bolus) after their baby is born.
  Interventions: Drug: Oxytocin
- 2 (Placebo Comparator): In one group, women will receive a small injection of saline (salt water) directly into the vein via their intravenous (bolus) after their baby is born.
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: Oxytocin — See detailed description
  Arms: 1
Drug: Saline solution — See detailed description
  Arms: 2

SUMMARY:
Oxytocin is normally given either rapidly into the vein (bolus) or put into an intravenous bag and administered more slowly, after delivery of the baby by cesarean section. Both of these methods are commonly used. To date there has been little research to demonstrate that one method of giving oxytocin is better than another in women who are more likely to bleed after delivery. The purpose of the study is to see whether a small bolus of oxytocin makes the uterus contract better to reduce bleeding and decreases the need to give additional oxytocin or more powerful drugs in women who are at risk for bleeding after delivery of their baby by cesarean section.

DETAILED DESCRIPTION:
Oxytocin is normally given either rapidly into the vein (bolus) or put into an intravenous bag and administered more slowly, after delivery of the baby by cesarean section. Both of these methods are commonly used. To date there has been little research to demonstrate that one method of giving oxytocin is better than another in women who are more likely to bleed after delivery. The purpose of the study is to see whether a small bolus of oxytocin makes the uterus contract better to reduce bleeding and decreases the need to give additional oxytocin or more powerful drugs in women who are at risk for bleeding after delivery of their baby by cesarean section.

Women who participate will be randomized (like a toss of a coin) to one of two groups. Neither the woman nor the anesthesiologist nor the obstetrician will know which group they are in.

In one group, the women will receive a small injection of saline (salt water) directly into the vein via their intravenous (bolus) after their baby is born. In the other group, the women will receive a small injection of oxytocin directly into the vein via their intravenous (bolus) after their baby is born.

Both groups will have the standard amount of oxytocin given slowly (over a 30 minute period) into the intravenous in their arm (infusion). The amount of oxytocin that is put into the intravenous bag is a normal amount that would be given during cesarean section in any woman not involved in the study and it will be started after the initial injection has been given. The only difference between the two groups is that one group will have an extra dose of oxytocin given directly into the vein via the intravenous while the other will have a saline solution given directly into the vein via the intravenous.

Information that will be obtained during the study will include any decrease in blood pressure or increase in heart rate at the time the saline or oxytocin is given directly into the vein. The obstetrician will be asked to indicate how well the uterus is contracting and they can ask the anesthesiologist to give more oxytocin or a more powerful drug if, in their opinion, the uterus is not contracting well. This is the normal way that this is done.

If the woman should feel dizzy (possibly secondary to low blood pressure) their anesthesiologist will treat them the same way as they would if this happened to any woman who is not part of the study. In other words, the anesthesiologist and obstetrician will treat the woman the way they normally would whether the woman was part of the study or not.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19 years or over
* Having a cesarean section
* Have one or more of the following

  1. a larger than average uterus, because of

     * a large baby
     * twins, triplets, etc
     * a large volume of fluid around the baby
  2. have received oxytocin to help stimulate labor for eight or more hours before cesarean section
  3. have infection inside the uterus that is treated with antibiotics
  4. bleeding after giving prior birth
  5. the placenta is in a position where it is more likely to bleed
  6. have had five or more pregnancies before current one

Exclusion Criteria:

* Significant medical problem such that an oxytocin bolus might not be safe
* Active bleeding and their blood pressure or pulse rate are not normal
* Blood does not clot normally
* Aged less than 19 years
* Does not understand English

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-11; Primary Completion 2006-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Need for additional oxytocics in women at high risk of hemorrhage | within the first hour after delivery

SECONDARY OUTCOMES:
Secondary outcomes include uterine tone and side effects. | within 10 minutes of delivery and time from giving the bolus until placenta delivery

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Douglas, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Department of Anesthesia, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] King KJ, Douglas MJ, Unger W, Wong A, King RA. Five unit bolus oxytocin at cesarean delivery in women at risk of atony: a randomized, double-blind, controlled trial. Anesth Analg. 2010 Dec;111(6):1460-6. doi: 10.1213/ANE.0b013e3181f8930a. Epub 2010 Oct 1. PMID 20889945